CLINICAL TRIAL: NCT04106999
Title: Dexmedetomidine and Inflammation in HIPEC Cases: A Case Series
Brief Title: Dexmedetomidine and HIPEC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jason Wilson, Clinical Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H19-00859
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Inflammation; Cancer
MeSH Terms: conditions — Inflammation; Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: 1 group will receive placebo drug delivery (Normal Saline infusion). The 2nd group will receive the study drug infusion (Dexmedetomidine)
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A blinded syringe with either the placebo or study drug will be given to the anesthesiologist involved in that patient's care. All other care providers will be blinded to the study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Normal Saline will be infused as per the protocol
  Interventions: Drug: Placebos
- Intervention group (Experimental): Dexmedetomidine will be infused as per the protocol
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Drug infusion will be delivered intra-operatively
  Arms: Intervention group
Drug: Placebos — Normal Saline will be infused as a control drug
  Arms: Placebo

SUMMARY:
Inflammation is associated with an increased risk of cancer recurrence. Various methods have been used to decrease the inflammatory response induced by the cancer and surgery. In this study the investigators would like determine if a commonly used sedative drug (dexmedtomidine) has an impact on this inflammatory state when used as part of the anesthetic. The investigators will conduct a pilot study with 20 patients undergoing a Hyperthermic Intraperitoneal Chemotherapy (HIPEC) procedure as part of their cancer treatment. 10 patients will receive the standard of care for anesthesia during the cancer surgery and a placebo infusion of normal saline at a rate consistent to that of the study drug. 10 additional patients will receive the same standard of care anesthetic plan with the addition of an infusion of dexmeditomidine during the procedure. The investigators will measure the degree of inflammation before, during and after the surgical procedure by looking at the levels of inflammatory markers in blood samples. The goal is to determine if the addition of dexmodtomidine affects the inflammatory state of patients undergoing a HIPEC procedure. This information will be used to guide future studies aiming at decreasing cancer recurrence and improve patient outcomes.

DETAILED DESCRIPTION:
Purpose: To investigate the use of intra-operative dexmedetomidine infusions to reduce the inflammatory and stress response of cytoreductive treatment and hyperthermic intra-peritoneal chemotherapy (HIPEC).

Hypothesis: HIPEC surgery patients who receive an intra-operative infusion of dexmedetomidine in addition to the current standard of care, consisting of parenteral and enteral opioids and thoracic epidural will have a reduction in their inflammatory markers intra-operatively, in PACU, POD1 and POD5 and a reduction in oral morphine equivalent opioid consumption in PACU and POD1, in comparison to those who receive a placebo infusion.

Justification: Surgical tumor excision is a cornerstone of primary cancer treatment, but is also recognized as one of the greatest risk factors for metastatic spread. The perioperative period, characterized by the surgical stress response and pharmacologic-induced angiogenesis and immunomodulation, results in a physiologic environment that supports tumor spread and distant reimplantation. There is potential for anesthesiologists to modulate the unwanted consequences of the stress response on the immune system and minimize residual disease by altering their anesthetic plan.

Dexmedtomidine is a commonly used sedative that can be used as part of an anesthetic during surgery. In vitro and animal studies have shown that dexmedtomidine decreases the inflammatory response but no research has been conducted with cancer-related conditions.

Objective: To determine if dexmedtomidine, when used intraoperatively, can decrease the levels of inflammation in patients a Hyperthermic Intraperitoneal Chemotherapy (HIPEC) procedure as part of their cancer treatment.

Primary Objective:

Reduction in inflammatory markers: CRP, ESR, NLR, PLR, plasma viscosity, lactate.

Secondary Objectives Reduction in Cancer markers: CEA (carcinoembyronic antigen] and CA19-9 Reduction in opioid use Reduction in volatile usage (average sevoflurane end-tidal level)

Research Design: In this pilot study, 20 patients undergoing a HIPEC procedure as part of their cancer treatment will be randomized into 2 groups. One group (controls) will receive the current anesthetic standard of care. The second group (experimental) will also receive the current anesthetic standard of care with the addition of an infusion of dexmedtomidine during the surgical procedure. Biomarkers of inflammation (Lactate, CRP, ESR, plasma viscosity, NLR, PLR, and procalcitonin) and cancer markers (CEA and CA19-9) will be measured at 5 time points: pre-operatively, intra-opertatively prior to chemotherapy, post-operatively in the post-anaesthetic care unit, post-operative day 1, and post-operative day 5. Quantitative analysis of the inflammatory markers will be used to compare the two groups.

Statistical Analysis: Data will be summarized and t-tests will be used to compare the data from the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a Hyperthermic Intraperitoneal Chemotherapy (HIPEC) procedure as part of their cancer treatment at Vancover General Hospital
* 18 years of age or older
* Able to provide informed consent
* Expected stay 5 days or greater in hospital
* Presenting for HIPEC with Colon or Appendix Cancer

Exclusion Criteria:

* Contraindication to dexmedtomidine use including allergy or sensitivity to the drug
* Pregnancy
* Dementia
* ASA greater than or equal to 4
* Significant liver disease
* Current use of steroid or immunosuppressive medication
* Mesothelioma tumour origin
* Current use of clonidine
* Current opioid use exceeding 30mg of oral morphine equivalents
* Patient not eligible or patient refusal to have a thoracic epidural

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Inflammation | 5 days
  Reduction in inflammatory markers: CRP, ESR, NLR, PLR, plasma viscosity, lactate.

SECONDARY OUTCOMES:
Cancer recurrance | 5 days
  Reduction in Cancer markers: CEA (carcinoembyronic antigen] and CA19-9
Anesthesia Dose | 5 days
  Reduction in volatile usage (average sevoflurane end-tidal level)
Opioid use | 5 days
  Reduction in opioid use

CONTACTS AND LOCATIONS:
Locations (1):
- UBC/Medicine, Faculty of/Anesthesiology, Pharmacology & Therapeutics, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We may publish this research and share at a conference or through a research paper